CLINICAL TRIAL: NCT04832243
Title: List Experiment to Measure Food and Water Insecurity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2013P000395_2
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Food Deprivation; Water Deprivation
Keywords: Food Insecurity; Water Insecurity
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Study participants are asked to identify the number of true statements in a list, where the number of true statements is randomly assigned. Neither study participants nor outcomes assessors are provided with information about "treatment" assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: V1: List No. 1 (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. The first version of the questionnaire includes 6 sets of 3 true-false statements that are innocuous and contextually applicable (e.g., weather, cultural norms) such that there is a low likelihood that the participant will answer untruthfully. The statements on food and water insecurity that are included in the experimental version are omitted.
  Interventions: Other: Survey questionnaire
- Experimental: V2: List No. 2 (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. The second version of the questionnaire includes 6 sets of 4 true-false statements that are innocuous and contextually applicable (e.g., weather, cultural norms) such that there is a low likelihood that the participant will answer untruthfully for 3 of the true-false statements. One statement in each set relates to food and water insecurity and is designed to determine the extent to which social desirability bias may influence responses to food and water insecurity questions.
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — Each version of the questionnaire includes a different number of true-false statements that study participants are asked to identify.

SUMMARY:
List experiment to measure food and water insecurity

DETAILED DESCRIPTION:
Food and water insecurity are complex, multi-domain constructs. Given their known association with important health and mental health outcomes, accurate assessment of food and water insecurity in resource-limited settings is paramount. The purpose of this study is to use a list experiment methodology to assess the extent to which there is bias in conventional survey-based means of direct elicitation of food and water insecurity. The list experiment provides an indirect means to measure a particular construct of interest. It is hypothesized that social desirability may cause upward bias in conventional survey-based means of direct elicitation of food and water insecurity.

ELIGIBILITY:
Inclusion Criteria:

* All adults who consider Nyakabare their primary place of residence and who are capable of providing consent

Exclusion Criteria:

* Minors younger than 18 years of age, with the exception of emancipated minors
* Persons who do not consider Nyakabare Parish their primary place of residence, e.g., persons who happen to be visiting Nyakabare at the time of the survey or who own a home in Nyakabare but spend most of their time outside the parish
* Persons with psychosis, neurological damage, acute intoxication, or other cognitive impairment (all of which are determined informally in the field by non-clinical research staff in consultation with a supervisor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1553 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
No Food Due to Lack of Money | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate even though participants are asked about the past month)
  "In the last month, was there ever no food to eat in the house because the participant lacked money to buy more?" (single item, culturally adapted from the 3-item Household Hunger Scale of USAID's Household Food Insecurity Access Scale [HFIAS]; response options yes/no)
No Water Due to Difficulty Collecting | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate even though participants are asked about the past month)
  "In the last month, was there ever no water in the participant's house because it was too difficult to collect more?" (single item, culturally adapted to indicate water insecurity, paralleling the 3-item Household Hunger Scale of USAID's Household Food Insecurity Access Scale [HFIAS]; response options yes/no)
Going to Sleep Hungry | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate even though participants are asked about the past month)
  "In the last month, did the participant or one of their household members ever go to sleep hungry because there was not enough food?" (single item, culturally adapted from the 3-item Household Hunger Scale of USAID's Household Food Insecurity Access Scale [HFIAS]; response options yes/no)
Going to Sleep Thirsty | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate even though participants are asked about the past month)
  "In the last month, did the participant or one of their household members ever go to sleep thirsty because there was not enough water?" (single item, culturally adapted to indicate water insecurity, paralleling the 3-item Household Hunger Scale of USAID's Household Food Insecurity Access Scale [HFIAS]; response options yes/no)
No Food for Entire Day | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate even though participants are asked about the past month)
  "In the last month, did the participant or one of their household members ever go an entire day and night without eating anything because there was not enough food?" (single item, culturally adapted from the 3-item Household Hunger Scale of USAID's Household Food Insecurity Access Scale [HFIAS]; response options yes/no)
Drink Unsafe Water | Baseline (The experimental manipulation in this study has to do with which version of the survey the study participant receives, so the time frame for assessment is immediate even though participants are asked about the past month)
  "In the last month, did the participant or one of their household members ever drink water that they thought might not be safe for their health?" (single item, culturally adapted to indicate water insecurity, developed specifically for this study; response options yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No